CLINICAL TRIAL: NCT06378138
Title: A Phase II/III Study of ICP-248 in Combination With Orelabrutinib in Patients With Treatment-naïve Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: ICP-248 in Combination With Orelabrutinib in Treatment-naïve Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (APEX-03)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01203
Record Dates: First submitted 2024-04-06; First posted 2024-04-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-248 in combination with Orelabrutinib (Experimental)
  Interventions: Drug: ICP-248; Drug: Orelabrutinib

INTERVENTIONS:
Drug: ICP-248 — Eligible patients will receive ICP-248 orally as per the protocol，once daily for every 28 days as one treatment cycle
Drug: Orelabrutinib — Eligible patients will receive Orelabrutinib orally as per the protocol，once daily for every 28 days as one treatment cycle

SUMMARY:
Evaluate the safety, tolerability and pharmacokinetics of ICP-248 in Combination with Orelabrutinib in Patients with Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years.
2. CLL/SLL is diagnosed by histopathology and/or flow cytometry according to the 2016 World Health Organization (WHO) classification criteria for lymphohematopoietic neoplasms or meeting the criteria of 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL 2018):
3. Having an indication for treatment that meets the criteria for iwCLL 2018
4. Subjects must have measurable lesion according to the Lugano 2014 Assessment Criteria.
5. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤ 2 and a life expectancy of ≥ 6 months.
6. Adequate hematologic function
7. Patients with basically normal coagulation function
8. Patients with adequate hepatic, renal, pulmonary and cardiac functions
9. Subjects are able to communicate with the investigator well and to complete the study as specified in the study.
10. Before the trial, the subjects shall understand the nature, significance, possible benefits, inconveniences and potential risks, as well as the study procedures of the trial in detail and voluntarily sign the written Informed Consent Form (ICF).

Exclusion Criteria:

1. Central nervous system involvement.
2. Concomitant Richter transformation.
3. Prior systemic treatment, excluding emergency pretreatment to reduce white blood cells and relieve leukostasis.
4. Requireing continuous glucocorticoid support or glucocorticoid therapy within 5 days.
5. History of allogeneic stem cell transplantation.
6. Major organ surgery (excluding aspiration biopsy) or significant trauma within 28 days prior to the first dose of the investigational drug or require elective surgery during the trial.
7. Presence of active infection that requires intravenous anti-infective therapy.
8. Hepatitis B or C virus infection.
9. History of immunodeficiency disease or Significant cardiovascular disease
10. Central nervous system disorders or Severe bleeding disorder
11. Alcohol or drug dependence.
12. Mental disorders or poor compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2030-11-25 (Estimated); Study Completion 2031-07-25 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) evaluation according to CTCAE V5.0 or iwCLL 2018 criteria | Up to 6 years
Changes from baseline in pulse. | Up to 6 years
Changes from baseline in blood pressure. | Up to 6 years
Changes from baseline in ECG QRS interval. | Up to 6 years
Changes from baseline in ECG QT interval. | Up to 6 years

CONTACTS AND LOCATIONS:
Locations (53):
- China (53):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital (The First Affiliated Hospital of University of Science and Technology of China), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, the Second Affiliated Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Affiliated Hospital of North China University of Science and Technology, Tangshan, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang City Center Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhenzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou First People's Hospital, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Bethune First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Linyi City Cancer Hospital, Linyi, Shandong
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Blood Diseases Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The People's Hospital Affiliated to Ningbo University, Ningbo, Zhejiang